CLINICAL TRIAL: NCT06929689
Title: Clinical and Radiographic Evaluation of All-on-three Immediately Loaded Mandibular Fixed Detachable Restorations (a Clinical Trial)
Brief Title: Evaluation of the All-on-three Concept in Mandible.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Naema Ammar, Assistant Lecturer at Removable Prosthodontics Department, Faculty of Dentistry, Pharos University, Alexandria, Egypt, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: all-on-three
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Dental Prosthesis; Dental Implant
Keywords: Three implants; Fixed detachable restorations

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- completely edentulous patients (Experimental): fixed detachable restorations on three dental implants in the mandible
  Interventions: Procedure: three dental implants

INTERVENTIONS:
Procedure: three dental implants — fixed detachable prosthesis

SUMMARY:
Evaluation of the clinical and radiographic treatment outcomes of immediately loaded three implants by fixed-detachable prostheses for the management of totally edentulous mandibles.

The hypothesis is that mandibular immediately loaded fixed detachable restorations supported only by three implants in the inter-foraminal region will not adversely affect the clinical or radiographical treatment outcome.

DETAILED DESCRIPTION:
The ideal amount of implants for edentulous mandible rehabilitation continues to be a subject of scholarly debate. Traditionally, at least four implants are required for fixed detachable prostheses, but increasing implant numbers raises costs and complexity, leading to patient reluctance. Reducing the number to three implants may simplify surgery, minimize trauma, and encourage patient acceptance.

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous patients with skeletal Class I maxilla-mandibular relationship.
* Adequate inter-arch space (22 mm), measured using the "try in" before any intervention.
* Male or female patients aged between 40 and 60 years.
* Maxillary and mandibular ridges with no history of recent extraction.
* Mandibular ridge should be ≥15 mm in height and ≥7 mm in width to accommodate three implants in the intra-foramina area of the mandibular arch, verified by using cone beam computed tomography (CBCT).

Exclusion Criteria:

* History of radiotherapy in the head and neck region.
* History of hard tissue augmentation.
* Presence of any intra-oral pathological condition.
* Any medical disorder that could complicate the surgical phase or affect osseointegration, such as osteoporosis, uncontrolled diabetes, and hypertension.
* Smoker and bruxer patients.

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-03-19 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2025-02-09 (Actual)

PRIMARY OUTCOMES:
Radiographic evaluation | 12 months
  The level of alveolar bone around each implant was evaluated using CBCT. Radiographic assessment of the vertical bone change around each implant was measured and the mean value was calculated. Bone measurements was evaluated at the insertion time then it was evaluated regularly 6 months and 12 months.
Peri-Implant Probing Depth (PIPD) | 12 months
  Peri-implant probing depth refers to the distance between the gingival margin and the most apically probable portion in millimeters (mm). The peri-implant sulcus depth was measured using a graduated plastic periodontal probe. The probe was held parallel to the long axis of the implant and introduced to the peri-implant sulcus with slight pressure. Measurements was made at four sites around each implant; buccal, lingual, mesial and distal. Probing depth of 1 mm or less was recorded as "1mm", and those exceeding 1 mm but less than 2 mm was recorded as "2mm" and so forth. The mean records for each implant was then calculated.
Clinical Attachment level (CAL) | 12 months
  It is the distance from the junction implant/abutment to the most apically probable portion, in millimeters. Assessment of the clinical attachment level was performed simultaneously while measuring the peri-implant probing depth.
Implant stability | 12 months
  Mobility (implant stability) was measured by using RFA (Osstell device instrument). The Osstell unit record numeric value of 1-100 which is referred to as the implant stability quotient (ISQ). The larger the ISQ value recorded indicates the more stable the implant-bone interface. Initial stability was checked at the insertion time then it was evaluated regularly, 6 months and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Abdelhamid, PhD, Study Chair — Alexandria University; Enaya Sharara, PhD, Study Chair — Alexandria University; Rania A Fahmy, PhD, Study Director — Alexandria University
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt